CLINICAL TRIAL: NCT00291759
Title: Adjuvant Endocrine Therapy in Postmenopausal Patients With HR +ve BC With Good to Moderate Differentiation - ARNO (Arimidex + Nolvadex). Primary Treatment for 2 Years With Tamoxifen Thereafter Randomisation to: Tamoxifen 3 Years or Anastrozole 3 Years.
Brief Title: ABCSG 8 - Adjuvant Treatment in Patients With Hormone Receptor-positive Breast Cancer With Good to Moderate Differentiation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1033AU/0002; ABCSG 8
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Anastrozole

INTERVENTIONS:
Drug: Tamoxifen
Drug: Anastrozole

SUMMARY:
The purpose of this study is to assess the difference in event-free survival between postmenopausal women with hormone receptor-positive early breast cancer who switched from tamoxifen to anastrozole and those who continued to receive tamoxifen.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mammary carcinoma after radical treatment, without prior chemo/hormone/radiation therapy.
* At least 6 lymph nodes examined.
* Good or intermediate tumour differentiation.
* <6 weeks before start of adjuvant therapy.
* Oestrogen or Progesterone positive

Exclusion Criteria:

* Premenopausal.
* Preoperative hormonal/antihormonal/radiation/cytoxic chemo. Second malignant tumour/status post second malignant tumour.
* In-situ/T4 carcinoma.
* Age >80 years.
* World Health Organisation performance index >3.
* Serious accompanying diseases

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3858 (Actual)
Dates: Start 1996-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To assess the difference in event free survival and overall survival (subject to stand-alone or combined/meta-analysis) between postmenopausal women with HR +ve early BC who switched from tamoxifen to anastrozole and those who continued on tamoxifen.

SECONDARY OUTCOMES:
To assess the difference in event free survival & overall survival (subject to stand-alone or combined/meta-analysis) plus side effects between postmenopausal women with HR+ve early BC who switched from tam to anastrozole and those who continued on tam.

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Jakesz, MD, Principal Investigator — Austrian Breast and Colorectal Cancer Study Group; AstraZeneca Austria Medical Director, MD, Study Director — AstraZeneca
Locations (52):
- Austria (52):
  - Research Site, Amstetten
  - Research Site, Bad Ischl
  - Research Site, Baden
  - Research Site, Bregenz
  - Research Site, Bruck/Mur
  - Research Site, Dornbirn
  - Research Site, Eisenstadt
  - Research Site, Feldbach
  - Research Site, Feldkirch
  - Research Site, Freistadt
  - Research Site, Fürstenfeld
  - Research Site, Gmünd
  - Research Sites, Graz
  - Research Site, Güssing
  - Research Site, Hainburg an der Donau
  - Research Site, Hartberg
  - Research Site, Hollabrunn
  - Research Site, Horn
  - Research Site, Innsbruck
  - Research Site, Judenburg
  - Research Site, Kirchdorf
  - Research Site, Klagenfurt
  - Research Sites, Klosterneuburg
  - Research Site, Kufstein
  - Research Site, Leoben
  - Research Sites, Linz
  - Research SIte, Melk
  - Research Site, Mistelbach
  - Research Site, Mödling
  - Research Site, Neunkirchen
  - Research Site, Oberpullendorf
  - Research Site, Oberwart
  - Research Site, Ried im Innkreis
  - Research Site, Rohrbach
  - Research Site, Rottenmann
  - Research Site, Saint Poelton
  - Research Site, Saint Veit/Glan
  - Research Site, Salzburg
  - Research Site, Schärding
  - Research Site, Scheibbs
  - Research Site, Schladming
  - Research Site, Schwarzach/Pongau
  - Research Site, Spittal/Drau
  - Research Site, Steyr
  - Research Site, Tulln
  - Research Sites, Vienna
  - Research Site, Villach
  - Research Site, Vöcklabruck
  - Research Site, Waidhofen/Thaya
  - Research Site, Wels
  - Research Site, Wolfsberg
  - Research Site, Zams

REFERENCES:
- [Derived] Sestak I, Cuzick J, Dowsett M, Lopez-Knowles E, Filipits M, Dubsky P, Cowens JW, Ferree S, Schaper C, Fesl C, Gnant M. Prediction of late distant recurrence after 5 years of endocrine treatment: a combined analysis of patients from the Austrian breast and colorectal cancer study group 8 and arimidex, tamoxifen alone or in combination randomized trials using the PAM50 risk of recurrence score. J Clin Oncol. 2015 Mar 10;33(8):916-22. doi: 10.1200/JCO.2014.55.6894. Epub 2014 Oct 20. PMID 25332252
- [Derived] Gnant M, Filipits M, Greil R, Stoeger H, Rudas M, Bago-Horvath Z, Mlineritsch B, Kwasny W, Knauer M, Singer C, Jakesz R, Dubsky P, Fitzal F, Bartsch R, Steger G, Balic M, Ressler S, Cowens JW, Storhoff J, Ferree S, Schaper C, Liu S, Fesl C, Nielsen TO; Austrian Breast and Colorectal Cancer Study Group. Predicting distant recurrence in receptor-positive breast cancer patients with limited clinicopathological risk: using the PAM50 Risk of Recurrence score in 1478 postmenopausal patients of the ABCSG-8 trial treated with adjuvant endocrine therapy alone. Ann Oncol. 2014 Feb;25(2):339-45. doi: 10.1093/annonc/mdt494. Epub 2013 Dec 16. PMID 24347518